CLINICAL TRIAL: NCT03631901
Title: Comparison Between Melatonin and Diazepam for Prevention of Recurrent Simple Febrile Seizures: Randomized Clinical Trial
Brief Title: Comparison Between Melatonin and Diazepam for Prevention of Recurrent Simple Febrile Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amira Hamed Darwish, Professor of pediatrics and Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TU2017
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Febrile Seizures
Keywords: Melatonin; Diazepam; recurrence; prophylaxis; Febrile convulsions
MeSH Terms: conditions — Seizures, Febrile; Recurrence | interventions — Melatonin; Diazepam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): melatonin 0.3mg/kg/8 hours, orally. Given only during the febrile illness.
  Interventions: Drug: oral melatonin
- Diazepam (Active Comparator): oral diazepam 1mg/kg/day divided into 3 doses. Given only during the febrile illness.
  Interventions: Drug: oral diazepam

INTERVENTIONS:
Drug: oral melatonin — Both melatonin and diazepam were given only during the febrile illness.
  Arms: Melatonin
Drug: oral diazepam — Both melatonin and diazepam were given only during the febrile illness.
  Arms: Diazepam

SUMMARY:
To evaluate the efficacy of oral melatonin compared to oral diazepam for prevention of recurrent simple febrile seizures.

DETAILED DESCRIPTION:
To evaluate the efficacy of oral melatonin compared to oral diazepam for prevention of recurrence of simple febrile seizures in children aged 6 months to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 5 yrs .
* Simple febrile seizures

Exclusion Criteria:

* Complex febrile seizures
* Child with history of neonatal seizure.
* Afebrile seizures.
* History of anticonvulsive therapy.
* Children suffering from epilepsy.
* Children with abnormal EEG.
* Children with abnormal neurological examination.
* Positive family history of epilepsy.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
recurrence of febrile seizures during febrile illness | 6 months

SECONDARY OUTCOMES:
side effect of medications reported in children | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amira Darwish, Principal Investigator — Tanta University Hospital
Locations (1):
- Tanta University, Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided